CLINICAL TRIAL: NCT01769638
Title: Safety and Pharmacokinetic Comparison of Sildenafil ODF and FCT Formulations in Healthy Korean Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0462
Record Dates: First submitted 2013-01-07; First posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
Keywords: Orally disintegrating Film; Film Coated Tablet; Sildenafil; Pharmacokinetics

ARMS (2):
- SPO1101 (Experimental)
  Interventions: Drug: SPO1101
- SPO1101D (Experimental)
  Interventions: Drug: SPO1101D

INTERVENTIONS:
Drug: SPO1101 — A single-dose of ODF and FCT formulations of sildenafil given orally in a fasted state (dose: 50mg), with a 7-day washout period between the formulations.
  Arms: SPO1101
Drug: SPO1101D — A single-dose of ODF and FCT formulations of sildenafil given orally in a fasted state (dose: 100mg), with a 7-day washout period between the formulations.
  Arms: SPO1101D

SUMMARY:
This study investigates safety and pharmacokinetic comparison of Seoul Pharma's orally disintegrating film (ODF) formulation of sildenafil (test formulation) and Pfizer's "Viagra® (sildenafil)" Film Coated Tablet (FCT) formulation (reference formulation) in healthy volunteers.

DETAILED DESCRIPTION:
* Background: An orally disintegrating film (ODF) formulation of sildenafil was recently developed in Korea. This formulation is expected to enhance the dosing convenience and increase patient compliance while yielding pharmacokinetic profiles comparable to the conventional film coated tablet (FCT) formulation.
* Objective: The goal of present study is to compare the pharmacokinetic (PK) profiles of a newly developed ODF formulation with a FCT formulation of sildenafil in healthy Korean male volunteers.
* Methods: This is a randomized, open-label, 2-period cross-over, single-dose study conducted in 2 parts. Eligible subjects were healthy male volunteers between the ages of 20 and 50 years and within 20% of their ideal body weight, and are equally divided into parts 1 and 2. Each subject will be received a single -dose of ODF and FCT formulations of sildenafil orally in a fasted state (part 1, 50mg; part 2, 100mg), with a 7-day washout period between the formulations. Blood samples are collected up to 24 hours. Pharmacokinetic parameters are determined for sildenafil and its active metabolite (N-desmethyl sildenafil). Adverse events will be also evaluated based on subject interviews and physical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were healthy male volunteers between the ages of 20 and 50 years and within 20% of their ideal body weight, and
* With no congenital abnormality or chronic disease.

Exclusion Criteria:

Key exclusion criteria included:

* history of cardiovascular, pulmonary, renal, endogenous, gastrointestinal, hematologic, neurologic, or hemorrhagic disease;
* anatomical abnormality of penis or factors that cause priapism (e.g., sicklemia, multiple myeloma, leukemia);
* clinically significant findings on routine laboratory (serology, hematology, serum chemistry, and urinalysis), ECG or color blindness tests [8, 16];
* history of hypersensitivity reaction to PDE5 inhibitor including sildenafil;
* use of prescription drugs within 14 days before the study that had the potential to interact with the study medication; and
* use of any substance that could induce or inhibit cytochrome P450 3A4 synthesis (eg, St. John's wort, other herbal medications).

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
AUC | 0 (predose), 0.017, 0.05, 0.117, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours after the dose

SECONDARY OUTCOMES:
Cmax | 0 (predose), 0.017, 0.05, 0.117, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours after the dose

REFERENCES:
- [Derived] Roh H, Son H, Lee D, Yeon KJ, Kim HS, Kim H, Park K. Pharmacokinetic comparison of an orally disintegrating film formulation with a film-coated tablet formulation of sildenafil in healthy Korean subjects: a randomized, open-label, single-dose, 2-period crossover study. Clin Ther. 2013 Mar;35(3):205-14. doi: 10.1016/j.clinthera.2013.02.006. PMID 23497759